CLINICAL TRIAL: NCT06927973
Title: Leveraging Exercise Stress Echocardiography for Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00117015
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-02

CONDITIONS: Chest Pain; Shortness of Breath
Keywords: Stress echocardiogram
MeSH Terms: conditions — Chest Pain; Dyspnea | interventions — Echocardiography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled subjects undergoing clinical stress echocardiogram (Experimental): The enrolled subject will undergo their clinically indicated stress echocardiogram study for chest pain or shortness of breath. At the conclusion of the clinical study 4 additional echo images will be obtained for research purposes.
  Interventions: Diagnostic Test: Echocardiogram

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Ultrasound

SUMMARY:
The purpose of this study is to find out if additional images taken during a stress echocardiogram study and risk score calculation will help the doctor determine if shortness of breath or chest pain are caused by stiff heart (heart failure with preserved ejection fraction or HFpEF).

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated exercise stress echo for the evaluation of exertional dyspnea or chest pain
* Age ≥50 years

Exclusion Criteria:

* Known history of HFpEF
* LVEF <50% on baseline echo study
* History of hypertrophic cardiomyopathy, amyloidosis, or pulmonary arterial hypertension, severe right ventricular dysfunction and severe valvular disease based on chart review or baseline echo study
* History of organ transplant (heart, kidney, liver, lungs)
* Severe pulmonary disease requiring ambulatory oxygen therapy
* End-stage renal disease requiring long-term renal replacement therapy
* Decompensated liver disease
* Conditions that prevent accurate assessment of E/e' ratio (mitral prosthetic valve, severe mitral annular calcification)
* Plan to use echo contrast agent during stress study (i.e. contrast agent needed for baseline study)
* Patients from outside Duke health system with no plan for long-term care at Duke

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
HFpEF clinic visit at 1 month and 6 months | Within 6 months of participant enrollment
  Number of participants undergoing resting only or exercise right heart catheterization
Confirmed HFpEF diagnosis at 1 month and 6 months | Within 6 months of participant enrollment
  Number of participants being documented to have HFpEF diagnosis in Electronic Health Record
Estimate the prevalence of undiagnosed HFpEF in patients undergoing exercise stress echo using HFpEF probability score and exercise echo filling pressure assessment | Within 6 months of participant enrollment
  Participants are presumed to have undiagnosed HFpEF using these following definitions:
  1. Participants with H2FPEF score ≥6
  2. Participants with elevated exercise echo filling pressure
  3. Participants with H2FPEF score ≥6 or elevated exercise echo filling pressure The difference in undiagnosed HFpEF prevalence between definition #1 and #3 will inform the incremental diagnostic value of exercise echo filling pressure assessment.

SECONDARY OUTCOMES:
Right heart catheterization (both resting and exercise) visit at 1 month and 6 months | Within 6 months of participant enrollment
  Number of participants undergoing resting only or exercise right heart catheterization
SGLT2 inhibitor use at baseline, months 1 and 6 | Baseline at enrollment and 6 months post enrollment
MRA Use at baseline, months 1 and 6 | Baseline at enrollment and 6 months post enrollment
GLP1 RA use at baseline, months 1 and 6 | Baseline at enrollment and 6 months post enrollment
Right heart catherization (both resting and exercise) referral at months 1 and 6 | Within 6 months of participant enrollment
HFpEF clinical referral at months 1 and 6 | Within 6 months of participant enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Marat Fudim, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No